CLINICAL TRIAL: NCT02305433
Title: Effects of Long-term Intensive Home-based Physiotherapy on Older People With an Operated Hip Fracture or Frailty (RCT).
Acronym: HIPFRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Karelia, Social and Health Care District (Other)
Collaborators: Social Insurance Institution, Finland (Other); University of Helsinki (Other); University of Jyvaskyla (Other); University of Eastern Finland (Other); University of Poitiers (Other); Ministry of Social Affairs and Health; Finland (Unknown)
Responsible Party: Principal Investigator, Paula Soukkio, Project Manager, South Karelia, Social and Health Care District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1236/00.01.05.01.00/2013
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Frail Elderly; Hip Fracture
Keywords: elderly; functional-based physiotherapy; frailty syndrome; osteoporotic hip fractures; home-based physiotherapy; home-dwelling; intervention; randomised controlled trial; costs of social and health care; quality of life; physical functioning; mobility; nutrition
MeSH Terms: conditions — Hip Fractures; Frailty | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physiotherapy (physical exercise) for frail elderly (Experimental): Individually tailored, long-term home-based physiotherapy (physical exercise)twice a week for 12 months. The duration of one session is 60 minutes.
  Interventions: Other: Home-based physiotherapy (physical exercise)
- Physiotherapy (physical exercise) for operated hip fracture patients (Experimental): Individually tailored, long-term home-based physiotherapy (physical exercise)twice a week for 12 months. The duration of one session is 60 minutes.
  Interventions: Other: Home-based physiotherapy (physical exercise)
- Usual care for frail elderly (No Intervention): Usual care follows the standard care procedures in the South Karelia Social and Health Care District in health care and in assisted home living.
- Usual care for operated hip fracture patients (No Intervention): Usual care follows the standard care procedures in the South Karelia Social and Health Care District in health care and in assisted home living.

INTERVENTIONS:
Other: Home-based physiotherapy (physical exercise) — Each physiotherapy (physical exercise) session includes muscle strength and endurance training (especially for lower limbs), balance and coordination training and functional training. Functional training includes walking exercises and ADL (activities of daily living) exercises. In addition the physiotherapist gives counseling on nutrition.
  Arms: Physiotherapy (physical exercise) for frail elderly; Physiotherapy (physical exercise) for operated hip fracture patients

SUMMARY:
Our objective is to study the effects of 12 months' intensive home-based physiotherapy (physical exercise) with 12 months' follow-up in two groups of older people: 1) those with an operated hip fracture (60+ y), and 2) those with signs of frailty (65+ y). The primary outcome measure is duration of living at home. Power calculations are based on the assumption that persons assigned to physiotherapy will live at home for six months longer vs. those in usual care. Secondary outcomes are physical functioning, falls, health-related quality-of-life, use and costs of social and health services, and mortality.

We will recruit 300 persons with hip fracture and 300 with signs of frailty in Eksote (South Karelia Social and Health Care District), Finland (population 133 000). The groups will be randomized separately into an intervention arm (home-based physiotherapy (physical exercise) twice a week for 12 months) and a control arm (usual care), resulting in 150 patients in each group.

An assessor-physiotherapist and assessor-nurse performs measurements at the participant's home at baseline, and after 3, 6 and 12 months. Assessments include, among others, Fried's frailty criteria, Short Physical Performance Battery (SPPB), Functional Independence Measure (FIM), Health-related quality-of-life (HRQoL, 15-D), Mini Nutritional Assessment (MNA), Falls Efficacy Scale - International (FES-I), Social Provision Scale (SPS), Mini Mental State Examination (MMSE), and Geriatric Depression Scale-15 (GDS-15). At 24 months we collect register information on mortality and the usage of health care services.

Recruitment will begin in December 2014 and last for three years. Data analyses and reporting will take place in 2017-21. The study is supported by the Social Insurance Institution of Finland, and the Ministry of Social Affairs and Health, Finland.

DETAILED DESCRIPTION:
There is increasing need to develop new models of rehabilitation to postpone older people's disabilities and institutional care. One alternative is home-based rehabilitation with emphasis on functional-based exercises and nutrition.

Our objective is to study the effects of home-based physiotherapy (physical exercise) for 12 months followed by 12 months' follow-up in older people, either with an operated hip fracture (60+ y) or with signs of frailty (65+ y). The primary outcome measure is duration of living at home (vs. assisted living and institutional care). Power calculations are based on the assumption that at 24 months persons assigned to physiotherapy (physical exercise) have lived at home for six months longer vs. those in usual care. Usual care follows the standard care procedures in South Karelia social and health care district (Eksote), Finland. The population in Eksote area is 133, 000. Secondary outcomes are physical functioning, falls, health-related quality-of-life (HRQoL), use and costs of social and health services, and mortality.

We will recruit 300 persons with hip fracture and 300 with signs of frailty. After the operation, persons with hip fracture will be transferred from the surgery unit to a rehabilitation hospital, where spend approximately four weeks before discharge. The other patient group includes persons with frailty signs. They will be screened among outpatients and inpatients using modified frailty questionnaires by Abellan van Kan et al. (2008) and Morley et al. (2012). Diagnosis of frailty is based on Fried´s criteria (2001). Both patient groups will be randomized separately into an intervention arm (home-based physiotherapy (physical exercise) twice a week for 12 months) and a control arm (usual care), resulting in 150 patients in each group.

Physiotherapy (physical exercise) is carried out by private physiotherapists, who have been trained to follow the intervention protocol. Physiotherapy (physical exercise) is individually designed to meet the patient's functional capacity and needs but at the same time it is progressive. Each physiotherapy (physical exercise) session includes muscle strength and endurance training (especially for lower limbs), balance and coordination training and functional training. Functional training includes activities of daily living (ADL) and walking exercises. In addition, the physiotherapists give counseling on nutrition (based on Mini Nutritional Assessment, MNA) and follow the participant´s weight.

An assessor-physiotherapist and assessor-nurse performs measurements at the participant's home at baseline, and after 3, 6 and 12 months. Assessments include, among others, modified Fried's frailty criteria, Short Physical Performance Battery (SPPB), Functional Independence Measure (FIM), HRQoL (15 D), MNA, Falls Efficacy Scale - International (FES-I), Social Provision Scale (SPS), Mini Mental State Examination (MMSE), and Geriatric Depression Scale-15 (GDS-15). In addition we collect register data on living and housing conditions, use and costs of social and health care services, and mortality at the end of the follow-up (24 months since the beginning of the study).

Recruitment will begin in December 2014 and last for three years. Data analyses and reporting will take place in 2017-21. The study is supported by the Social Insurance Institution of Finland, and the Ministry of Social Affairs and Health, Finland.

References

* Abellan van Kan G, Rolland Y, Bergman H, Morley JE, Kritchevsky SB, Vellas B. (2008). The I.A.N.A Task Force on frailty assessment of older people in clinical practice. J Nutr Health Aging.12(1):29-37
* Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA. (2001). Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci;56(3):M146-56.
* Morley JE, Malmstrom TK, Miller DK.(2012). A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging 16(7):601-8.

ELIGIBILITY:
Inclusion Criteria:

* age 65+ for frail persons and 60 + for hip fracture patients
* home-dwelling but an increased risk for disabilities or for institutional care
* ability to walk inside one´s own home with or without mobility aids
* ability to communicate in Finnish
* in case of hip fracture: the first operated hip fracture
* in case of frailty: signs of frailty assessed by modified Fried's frailty criteria

Exclusion Criteria:

* living in nursing home or institutional care facility
* severe neurological diseases (Parkinson, MS, stroke)
* severe heart diseases with physical capacities significantly impaired (NYHA class III or IV)
* severe musculoskeletal diseases which prevent from participating in long-term physiotherapy
* terminal illnesses (e.g. cancer) that diminish the estimated home-dwelling time to less than two years
* severe mental problems (severe depression, psychosis or schizophrenia)
* severe alcohol or drug abuse
* severe problems with hearing or eyesight

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2014-12; Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
duration of time living at home | 24 months
  register information

SECONDARY OUTCOMES:
change in physical functioning | baseline and 3, 6, 12 months
  Short Physical Performance Battery, Hand grip strength, Functional Independence Measure, Instrumental Activities of Daily Living, physical activity
the amount of use of social and health services | baseline and 12 and 24 months
  register information, the amount of primary and secondary healthcare and social services used during study period (two years) gathered from the electronic medical records
the cost of the social and health services used | baseline and 12 and 24 months
  register information, the amount of services calculated by multiplying the number of service units used with the national mean unit costs
change in health-related quality-of-life | baseline and 3, 6, 12 months
  15D© which has fifteen items, each having five answer options, A set of utility or preference weights is used to generate the 15D score (single index number) on a 0-1 scale (1=full health, 0=death).
change in severity of frailty | baseline and 12 months
  modified Fried´s frailty criteria
all cause mortality | 3, 6, 12 and 24 months
  register information
the amount of falls | baseline and 3, 6, 12 months
  diary, register information

CONTACTS AND LOCATIONS:
Overall Officials: Markku T Hupli, MD, PhD, Study Director — Treenix
Locations (1):
- South Karelia Social and Health Care District, Lappeenranta, South Karelia Region, Finland

IPD SHARING:
Plan to Share IPD: No
This was not planned in advance in the original study plan. We do not have participants permission to share our data.

REFERENCES:
- [Background] Soukkio P, Suikkanen S, Kaaria S, Kautiainen H, Sipila S, Kukkonen-Harjula K, Hupli M. Effects of 12-month home-based physiotherapy on duration of living at home and functional capacity among older persons with signs of frailty or with a recent hip fracture - protocol of a randomized controlled trial (HIPFRA study). BMC Geriatr. 2018 Oct 1;18(1):232. doi: 10.1186/s12877-018-0916-y. PMID 30285645
- [Result] Soukkio PK, Suikkanen SA, Aartolahti EM, Kautiainen H, Kaaria SM, Hupli MT, Pitkala KH, Sipila S, Kukkonen-Harjula KT. Effects of Home-Based Physical Exercise on Days at Home, Health Care Utilization, and Functional Independence Among Patients With Hip Fractures: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Sep;102(9):1692-1699. doi: 10.1016/j.apmr.2021.04.004. Epub 2021 Apr 30. PMID 33939973
- [Result] Soukkio PK, Suikkanen SA, Kukkonen-Harjula KT, Kautiainen H, Hupli MT, Aartolahti EM, Kaaria SM, Pitkala KH, Sipila S. Effects of a 12-month home-based exercise program on functioning after hip fracture - Secondary analyses of an RCT. J Am Geriatr Soc. 2022 Sep;70(9):2561-2570. doi: 10.1111/jgs.17824. Epub 2022 May 18. PMID 35582993
- [Result] Suikkanen S, Soukkio P, Pitkala K, Kaaria S, Kautiainen H, Sipila S, Kukkonen-Harjula K, Hupli M. Older persons with signs of frailty in a home-based physical exercise intervention: baseline characteristics of an RCT. Aging Clin Exp Res. 2019 Oct;31(10):1419-1427. doi: 10.1007/s40520-019-01180-z. Epub 2019 Apr 2. PMID 30941731
- [Result] Suikkanen SA, Soukkio PK, Aartolahti EM, Kautiainen H, Kaaria SM, Hupli MT, Sipila S, Pitkala KH, Kukkonen-Harjula KT. Effects of Home-Based Physical Exercise on Days at Home and Cost-Effectiveness in Pre-Frail and Frail Persons: Randomized Controlled Trial. J Am Med Dir Assoc. 2021 Apr;22(4):773-779. doi: 10.1016/j.jamda.2020.06.005. Epub 2020 Jul 18. PMID 32694001
- [Result] Suikkanen S, Soukkio P, Aartolahti E, Kaaria S, Kautiainen H, Hupli MT, Pitkala K, Sipila S, Kukkonen-Harjula K. Effect of 12-Month Supervised, Home-Based Physical Exercise on Functioning Among Persons With Signs of Frailty: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Dec;102(12):2283-2290. doi: 10.1016/j.apmr.2021.06.017. Epub 2021 Jul 18. PMID 34283997
- [Result] Suikkanen S, Soukkio P, Kautiainen H, Kaaria S, Hupli MT, Sipila S, Pitkala K, Aartolahti E, Kukkonen-Harjula K. Changes in the Severity of Frailty Among Older Adults After 12 Months of Supervised Home-Based Physical Exercise: A Randomized Clinical Trial. J Am Med Dir Assoc. 2022 Oct;23(10):1717.e9-1717.e15. doi: 10.1016/j.jamda.2022.07.010. Epub 2022 Aug 18. PMID 35985418
- [Derived] Suikkanen S, Soukkio P, Kantola M, Kautiainen H, Haanpaa M, Hupli MT, Kukkonen-Harjula K. Long-term home-based physical exercise, pain, and use of pain medication over a year after hip fracture - A secondary analysis of a randomised controlled trial. Clin Rehabil. 2026 Feb;40(2):193-206. doi: 10.1177/02692155251389435. Epub 2025 Oct 23. PMID 41130912
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- See also: The study report of the results of other secondary outcomes in Finnish. — http://urn.fi/URN:NBN:fi-fe2022091459015
- See also: The study protocol and details of the intervention and participating in the intervntion in Finnish. — http://urn.fi/URN:NBN:fi-fe202001233112
- See also: PhD thesis, Sara Suikkanen: Home-Based Physical Exercise Among Older Adults with Signs of Frailty - Emphasis on Days Lived at Home, Utilization of Social and Health Care Services, Quality of Life, Physical Functioning, and Severity of Frailty — https://jyx.jyu.fi/handle/123456789/84173